CLINICAL TRIAL: NCT03991533
Title: Use of Multiparametric Magnetic Resonance Imaging in the Management of Head and Neck Cancer
Brief Title: Use of Multiparametric MRI in the Management of Head and Neck Cancer: a Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, Principal investigator, AZ Sint-Jan AV
Other Study IDs: 2360
Record Dates: First submitted 2019-02-13; First posted 2019-06-19 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer; Multiparametric MRI; Cervical Lymph Node
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- affected: patients with a histologically confirmed head and neck tumour
  Interventions: Other: multiparametric MRI
- control: histologically confirmed Whartin tumour or pleomorphic adenoma of the parotid gland, without malignant transformation
  Interventions: Other: multiparametric MRI

INTERVENTIONS:
Other: multiparametric MRI — preoperative multiparametric MRI

SUMMARY:
The investigators aim to identify specific MRI parameters that could improve diagnostic accuracy of metastatic cervical lymph nodes in patients with a squamous cell carcinoma in the head and neck region.

DETAILED DESCRIPTION:
Background:The locoregional control rates in patients with advanced head and neck cancer remain suboptimal. Accurate diagnosis of metastatic cervical lymph nodes remains challenging. Technological advances in magnetic resonance imaging (MRI) enable to quantify diffusion and perfusion of the tumour and its surrounding tissues, which could improve diagnostic performance.

Objectives: The investigators aim to identify specific MRI parameters that could improve diagnostic accuracy of metastatic cervical lymph nodes in patients with a squamous cell carcinoma in the head and neck region.

Study design: a retrospective study will be set up to explore the diagnostic performance of the selected MRI parameters to differentiate between tumoural and non-tumoural cervical lymph nodes in patients with a histologically confirmed head and neck tumour ('affected group') or histologically confirmed Whartin tumour or pleomorphic adenoma of the parotid gland, without malignant transformation ('control group').

Patients will be screened for inclusion in the analysis if they had a routine preoperative multiparametric MRI, according to a standardised protocol, between the 1st of December 2016 and the 30th of September 2018. All MR images will be screened by the resident to select those patients with one or multiple clearly distinguishable metastatic cervical lymph node(s), which can be clearly correlated with the final pathology report. Other strict inclusion criteria are described in detail in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* patients that received a pretreatment multiparametric MRI according to a standardized protocol between December 2016 and December 2018
* histophatologically proven SCC in the head and neck region
* one or multiple clearly distinguishable cervical lymph node(s), that can be unambiguously correlated with the pathology report

Exclusion Criteria:

* patients not fulfilling abovementioned criteria
* patients with thyroid or skin cancer
* considerable artefact on MRI
* previous surgery, irradiation or chemotherapy in the HN region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: affected group: Histopathologically proven SCC in the HN region control group: Histopathologically proven Whartin tumour or pleomorphic adenoma of the parotid gland, without malignant transformation in the HN region
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
discriminatory value of MRI perfusion curve | preoperative
  differentiation between a metastatic cervical lymph node and a non-tumoural lymph node, as based on the final pathology report as the 'gold standard'
discriminatory value of MRI ADC | preoperative
  differentiation between a metastatic cervical lymph node and a non-tumoural lymph node, as based on the final pathology report as the 'gold standard'
discriminatory value of MRI D-value | preoperative
  differentiation between a metastatic cervical lymph node and a non-tumoural lymph node, as based on the final pathology report as the 'gold standard'

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — AZ Sint-Lucas Brugge

IPD SHARING:
Plan to Share IPD: No